CLINICAL TRIAL: NCT01857973
Title: In-Clinic Feasibility Study to Observe the Overnight Closed Loop System
Brief Title: Overnight Closed Loop Study in U.S.
Acronym: OCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CEP273
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes
Keywords: HCL; Type 1 Diabetes; Sensor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: subjects undergo treatment with the hybrid closed loop system under various experimental conditions
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hybrid Closed Loop (Experimental): In-clinic evaluation of the HCL System under various conditions.
  Interventions: Device: Hybrid Closed Loop

INTERVENTIONS:
Device: Hybrid Closed Loop — The Hybrid Closed Loop System is an investigational device intended for closed loop control of blood glucose.

SUMMARY:
This is a multicenter feasibility study. Up to 85 subjects will be enrolled in the study. The goal of the study is to demonstrate that the Hybrid Closed Loop (HCL) System is safe to be used in an even larger study outside of hospital.

DETAILED DESCRIPTION:
Subjects that have met eligibility criteria will undergo treatment with the hybrid closed loop system under various experimental conditions.There is no statistically powered study hypothesis testing.

The investigational centers will be encouraged to include subjects of different ethnicities including Hispanic, Native American, and African-American.

The study is anticipated to last no more than 12 months from investigational center initiation to finalization of all data entry and monitoring procedures. Subjects are expected to participate for approximately 1- 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 2-75 years of age at time of screening
2. A clinical diagnosis of type 1 diabetes as determined by either medical record or source documentation from qualified individual to make medical diagnosis

   Exclusion Criteria that are Based on Demands of In-Clinic Study Procedures :
3. Pump therapy for greater than 6 months with use of real time CGM for any period of time (ie. one day) 3 months prior to screening
4. Adequate venous access as assessed by investigator or appropriate staff
5. Subject should have an established insulin carbohydrate and insulin sensitivity ratio.
6. Subject reports at the time of screening that their average fasting glucose is 60 mg/dL - 200 mg/dL
7. Subject reports at the time of screening that their average total daily insulin dose is 15 units - 110 units. (Insulin pump memory for this information may be used)

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lee, MD, Study Director — Medtronic
Locations (6):
- United States (6):
  - AMCR Institute, Inc. 700 West El Norte Parkway, Suite 201, Escondido, California
  - Barbara Davis Center, 1775 Aurora Court, A140, Aurora, Colorado
  - Yale University School of Medicine, 2 Church Street South, Suite 404, New Haven, Connecticut
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - University of Virginia, 617 West Main Street, 4th Floor, Charlottesville, Virginia
  - Rainier Clinical Research, 723 SW 10th Street, Suite 100, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 phases: Exploratory A, Exploratory B, Phase 1, Phase 2, Phase 3, Phase 4, Phase 6 and Phase 7.
Period: Overall Study
Arm/Group | Hybrid Closed Loop
Started | 78
Exploratory A Phase | 9
Xploratory B Phase | 9
Phase 1 | 17
Phase 2 | 14
Phase 3 | 10
Phase 4 | 10
Phase 6 | 4
Phase 7 | 4
Completed | 73
Not Completed | 5
Not completed — Subject did not meet required BG range | 3
Not completed — drop out after 3 failed attempts | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (16.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Euglycemic Range - Phase 3 (Closed-loop Using the NGP Pump Platform)
Description: time in euglycemic range (% of Senosr Glucose (SG) 70-180 mg/dL), Phase 3 (closed-loop using the Next Generation Pump (NGP) platform). The experiment was conducted in a monitored setting which lasted for 12 days with the following stressors: missed meal bolus, exercise, missed transmission, Umax (maximum insulin limit) challenges. The study was conducted in a clinic or hotel/house environment for 12 days/11 nights with no dietary or activity restrictions.
Time Frame: 12 days
Population: Eight type-1 diabetic subjects participated in this phase.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 8
percentage of time | 69.3 (8.9)

2. Secondary Outcome: Percentage of Time in Euglycemic Range - Exploratory A Phase
Description: Percentage of time in euglycemic range (% of SG 70-180 mg/dL) - Exploratory A phase. An overnight closed-loop experiment was performed using the Android Development Platform, software version 2.0 A system's closed-loop algorithm without implementing the upper-limit for insulin delivery.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 8
percentage of time | 90.7 (13.3)

3. Secondary Outcome: Number of Subject With YSI (Yellow Spring Instrument) Dipped Below 50mg/dL - Exploratory B Phase
Description: The purpose of exploratory B study was to evaluate the efficacy and safety of the insulin upper-limit, Umax. The Umax is a patient-specific parameter which is calculated based on historical data from the pump that includes SG tracings, insulin delivery information, and the carbohydrate inputs from the user. The main objective of Umax is to prevent the user from being severely hypoglycemic (less than 50 mg/dL) by restricting the controller from over-delivery of insulin.
Time Frame: 1 day
Population: Five out of the eight subjects with YSI dipped below 50mg/dL
Measure: Number; unit: number of subjects
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 8
number of subjects | 5

4. Secondary Outcome: Number of Subject Under-calibrated to Introduce a Persistent Under-reading Sensor Measurement Bias- Phase 1
Description: Number of subject under-calibrated to introduce a persistent under-reading sensor measurement bias- Phase 1
Time Frame: 1 day
Population: 13 subjects with sensors under-calibrated to introduce a persistent under-reading sensor measurement bias
Measure: Number; unit: participants
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 16
participants | 13

5. Secondary Outcome: Percentage of Time in Euglycemic Range - Phase 2
Description: Percentage of time in euglycemic range (% of SG 70-180 mg/dL) - Phase 2
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 14
percentage of time | 65.8 (16.2)

6. Secondary Outcome: Percentage of Time in Euglycemic Range - Phase 4
Description: Percentage of time in euglycemic range (% of SG 70-180 mg/dL) - Phase 4
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 10
percentage of time | 76.1 (8.6)

7. Secondary Outcome: Percentage of Time in Euglycemic Range - Phase 6
Description: Percentage of time in euglycemic range (% of SG 70-180 mg/dL) - Phase 6
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 4
percentage of time | 60 (8.0)

8. Secondary Outcome: Percentage of Time in Euglycemic Range - Phase 7
Description: Percentage of time in euglycemic range (% of SG 70-180 mg/dL) - Phase 7
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Hybrid Closed Loop
Number analyzed (Participants) | 4
percentage of time | 60 (24.9)

ADVERSE EVENTS:
Time Frame: 30 - 60 days
Arm/Group | Hybrid Closed Loop
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 7/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid Closed Loop (N=78)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left arm pain due to IV placement (General disorders) | 1 (1)
Right arm pain due to IV placement (General disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial petechiae of the eyes (Skin and subcutaneous tissue disorders) | 1 (1)
costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Common cold (Infections and infestations) | 1 (1)
Severe hyperglycemia (Metabolism and nutrition disorders) | 1 (4)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days